CLINICAL TRIAL: NCT00119678
Title: A Phase IIB, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Abatacept vs Placebo on a Background of Oral Glucocorticosteroids in the Treatment of Subjects With Systemic Lupus Erythematosus and the Prevention of Subsequent Lupus Flares
Brief Title: Abatacept in the Treatment and Prevention of Active Systemic Lupus Erythematosus (SLE) Flares in Combination With Prednisone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IM101-042
Record Dates: First submitted 2005-06-30; First posted 2005-07-14 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Abatacept; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abatacept + Prednisone (Active Comparator): Double Blind Period
  Interventions: Drug: Abatacept; Drug: Prednisone
- Placebo + Prednisone (Placebo Comparator): Double Blind Period
  Interventions: Drug: Placebo; Drug: Prednisone
- Abatacept (Experimental): Open Label
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Injectable, intravenous, 10 mg/kg, abatacept every 28 days, 12 months
  Other Names: Orencia
  Arms: Abatacept + Prednisone
Drug: Placebo — Injectable, intravenous, 0 mg, every 28 days, 12 months
  Arms: Placebo + Prednisone
Drug: Prednisone — Tablets, oral, 30 mg, daily for 28 days then taper off, 12 months
  Arms: Abatacept + Prednisone; Placebo + Prednisone
Drug: Abatacept — Injectable, intravenous, 10 mg/kg, every 28 days
  Other Names: Orencia
  Arms: Abatacept

SUMMARY:
The purpose of this clinical research study is to learn whether Abatacept can treat and prevent lupus flares; specifically, in patients with active lupus flares in at least one of three organ systems: skin (discoid lesions); inflammation of the lining of the heart (pericarditis), or inflammation of the lining of the lung (pleuritis/pleurisy); or inflammation of more than 4 joints (arthritis). All participants will receive prednisone or prednisone-equivalent treatment in combination with study medication. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* participants must be diagnosed with SLE and be experiencing an active lupus flare in at least one of three organ systems: skin (discoid lesions), inflammation of the lining of the heart (pericarditis), or inflammation of the lining of the lung (pleuritis/pleurisy); or inflammation of more than 4 joints within 14 days of a screening visit (arthritis)
* Stable dose of prednisone (<30mg) for at least one month

Exclusion Criteria:

* participants experiencing an active lupus flare in the kidney or central nervous systems
* Treatment with a stable dose of azathioprine, mycophenolate mofetil, hydroxychloroquine, chloroquine, or methotrexate for less than three months prior to the study
* participants with active viral or bacterial infections
* participants with any other autoimmune disease as a main diagnosis
* Prior treatment with rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (46):
- United States (12):
  - University Of Arizona Arthritis Center, Tucson, Arizona
  - Office Of Geoffrey S. Dolan, Md, Long Beach, California
  - 8737 Beverly Blvd., Los Angeles, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Cria Research, Fort Lauderdale, Florida
  - The University Of Chicago, Chicago, Illinois
  - Kentuckiana Center For Better Bone And Joint Health, Louisville, Kentucky
  - Kelly, Timothy, Las Vegas, Nevada
  - Suny Downstate Medical Center, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Ok Medical Research Foundations, Oklahoma City, Oklahoma
  - Texas Research Center, Sugarland, Texas
- Australia (5):
  - Local Institution, Cairns, Queensland
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Clayton, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Malvern, Victoria
- Local Institution, Graz, Austria
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Brazil (5):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro - Rj, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (2):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
- France (3):
  - Local Institution, Bordeaux
  - Local Institution, Montpellier
  - Local Institution, Paris
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Düsseldorf
  - Local Institution, Freiburg im Breisgau
- Local Institution, Ferrara, Italy
- Mexico (3):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michioacan
- Local Institution, Ponce, Puerto Rico
- South Africa (2):
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
- South Korea (2):
  - Local Institution, Seoul, Sungdong-Gu
  - Local Institution, Seoul
- Taiwan (3):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taipei
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Hu Y, Carman JA, Holloway D, Kansal S, Fan L, Goldstine C, Lee D, Somerville JE, Latek R, Townsend R, Johnsen A, Connolly S, Bandyopadhyay S, Shadick N, Weinblatt ME, Furie R, Nadler SG. Development of a Molecular Signature to Monitor Pharmacodynamic Responses Mediated by In Vivo Administration of Glucocorticoids. Arthritis Rheumatol. 2018 Aug;70(8):1331-1342. doi: 10.1002/art.40476. Epub 2018 Jul 12. PMID 29534336
- [Derived] Bandyopadhyay S, Connolly SE, Jabado O, Ye J, Kelly S, Maldonado MA, Westhovens R, Nash P, Merrill JT, Townsend RM. Identification of biomarkers of response to abatacept in patients with SLE using deconvolution of whole blood transcriptomic data from a phase IIb clinical trial. Lupus Sci Med. 2017 Jul 28;4(1):e000206. doi: 10.1136/lupus-2017-000206. eCollection 2017. PMID 29214034
- [Derived] Merrill JT, Burgos-Vargas R, Westhovens R, Chalmers A, D'Cruz D, Wallace DJ, Bae SC, Sigal L, Becker JC, Kelly S, Raghupathi K, Li T, Peng Y, Kinaszczuk M, Nash P. The efficacy and safety of abatacept in patients with non-life-threatening manifestations of systemic lupus erythematosus: results of a twelve-month, multicenter, exploratory, phase IIb, randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2010 Oct;62(10):3077-87. doi: 10.1002/art.27601. PMID 20533545

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 263 participants were enrolled in this study and 80 were excluded from the trial due to screening failure. Of the 183 randomized, 3 were not treated and 5 were treated but excluded due to site closure.
Groups:
- Abatacept: Participants were administered intravenous (iv) infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 337. All participants received a dose based on screening visit weight. Prednisone or prednisone equivalent was administered at an initial oral dose of 30 mg once daily (OD). A standardized prednisone or prednisone equivalent taper procedure was followed whenever the participant's clinical features qualified for British Isles Lupus Assessment Group (BILAG) "C" or "D" status after Day 29. Participants who completed the double-blind period were eligible for the open-label long-term extension period, where all participants were reallocated to abatacept (regardless of randomized treatment in the double-blind period) according to body weight at study entry. Infusions continued every 28 days until abatacept was marketed for SLE or the drug development program discontinued.
- Placebo: Participants were administered iv infusions of either dextrose 5% solution or normal saline (NS) at a constant rate over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 337. Prednisone or prednisone equivalent was administered at an initial oral dose of 30 mg OD. A standardized prednisone or prednisone equivalent taper procedure was followed whenever the participant's clinical features qualified for BILAG "C" or "D" status after Day 29. Participants who completed the double-blind period were eligible for the open-label long-term extension period, where all participants were reallocated to abatacept (regardless of randomized treatment in the double-blind period) according to body weight at study entry. Infusions continued every 28 days until abatacept was marketed for SLE or the drug development program discontinued.
Period: Double-blind Treatment Period
Arm/Group | Abatacept | Placebo
Started | 122 | 61
RANDOMIZED AND TREATED | 121 | 59
RANDOMIZED,TREATED, AND ANALYZED | 118 | 57
Completed | 81 | 35
Not Completed | 41 | 26
Not completed — Death | 1 | 0
Not completed — Adverse Event | 7 | 1
Not completed — Lack of Efficacy | 21 | 12
Not completed — Lost to Follow-up | 1 | 2
Not completed — Participant withdrew consent | 4 | 4
Not completed — Participants not meeting study criteria | 0 | 1
Not completed — Poor/Non-compliance | 3 | 0
Not completed — Pregnancy | 0 | 2
Not completed — Not treated | 1 | 2
Not completed — Site closed due to non-compliance | 3 | 2
Period: Open-label Treatment Period
Arm/Group | Abatacept | Placebo
Started | 110 (Number of participants treated) | 0
Completed | 0 | 0
Not Completed | 110 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 9 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Participant withdrew consent | 4 | 0
Not completed — Participants not meeting study criteria | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Administrative reasons by sponsor | 87 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 118 | 57 | 175
Age, Continuous [Median (Full Range); unit: years] — 183 participants were randomized, 3 were not treated and 5 were treated but excluded due to site closure. Thus, Abatacept group n=118 and Placebo group n=57.
  years | 38.0 (12.76) [18.0 to 71.0] | 36.0 [19.0 to 65.0] | 38.0 [18.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants] — 183 participants were randomized, 3 were not treated and 5 were treated but excluded due to site closure. Thus, Abatacept group n=118 and Placebo group n=57.
  Participants
    Female | 104 | 55 | 159
    Male | 14 | 2 | 16
Race/Ethnicity, Customized [Number; unit: participants] — 183 participants were randomized, 3 were not treated and 5 were treated but excluded due to site closure. Thus, Abatacept group n=118 and Placebo group n=57.
  participants
    White | 74 | 39 | 113
    Black/African American | 12 | 4 | 16
    American Indian/Alaska Native | 1 | 0 | 1
    Asian | 28 | 13 | 41
    Other races | 3 | 1 | 4
Weight [Mean (Standard Deviation); unit: kilograms] — 183 participants were randomized, 3 were not treated and 5 were treated but excluded due to site closure. Thus, Abatacept group n=118 and Placebo group n=57.
  kilograms | 68.630 (18.717) | 69.000 (14.790) | 68.750 (17.493)
Systemic Lupus International Collaborative Clinics/American College of Rheumatology(SLICC/ACC) score [Number; unit: participants] — SLICC/ACR score or damage index is a measure of cumulative damage due to Systemic Lupus Erythematosus (SLE). Damage is defined as non-reversible change (not related to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months. A score of 0=no damage, early damage is defined as ≥1. The total maximum score is 48, and increasing score indicates increasing disease severity. 183 participants were randomized, 3 were not treated and 5 were treated but excluded due to site closure. Thus, Abatacept group n=118 and Placebo group n=57.
  participants
    Overall SLICC/ACR score 0 | 82 | 38 | 120
    Overall SLICC/ACR score 1 | 12 | 11 | 23
    Overall SLICC/ACR score 2 | 15 | 5 | 20
    Overall SLICC/ACR score >2 | 6 | 1 | 7
    Overall SLICC/ACR score unavailable | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Period (DB); Number of Participants Experiencing a New SLE Flare
Description: SLE flares scored using BILAG:A:presence of =>1 serious;B:more moderate;C:mild symptomatic;D:prior activity,no current symptoms;E:organ that has never been involved. Calculated based on change during previous 4 weeks (1=improving,2=staying same,3=worsening,4=new).New SLE flare:first BILAG 'A' or 'B' event adjudicated to be flare following resolution of entry flare and start of prednisone/prednisone-equivalent taper.Inception treatment failure included (entry flare did not subside by Day 57/participant discontinued double-blind period before Day 29).
Time Frame: From start of corticosteroid taper to Day 365
Population: All randomized and treated participants, grouped by the treatment randomized to (Intent to Treat [ITT]). Participants who were inception treatment failures were treated as having 1 new flare; participants who discontinued early without any new flares were treated as having 1 new flare.
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 118 | 57
Participants | 94 [72.4 to 86.9] | 47 [72.6 to 92.3]

2. Secondary Outcome: DB; Number of Participants With a New SLE Flare During the Initial 6 Months
Description: SLE flares scored using BILAG:A:presence of =>1 serious;B:more moderate;C:mild symptomatic;D:prior activity,no current symptoms;E:organ that has never been involved.Calculated based on change during previous 4 weeks (1=improving,2=staying same,3=worsening,4=new).New SLE flare:first BILAG 'A' or 'B' event adjudicated to be flare following resolution of entry flare and/or start of prednisone/prednisone-equivalent taper.Inception treatment failure included (entry flare did not subside by Day 57/participant discontinued double-blind period before Day 29).
Time Frame: From start of corticosteroid taper to 6 months.
Population: All randomized and treated participants, grouped by the treatment randomized to (ITT).
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 118 | 57
Participants | 75 [54.9 to 72.2] | 36 [50.6 to 75.7]

3. Secondary Outcome: DB; Total Number of New SLE Flares Each Participant Experienced
Description: SLE flares scored using BILAG:A:presence of =>1 serious;B:more moderate;C:mild symptomatic;D:prior activity,no current symptoms;E:organ that has never been involved.Calculated based on change during previous 4 weeks (1=improving,2=staying same,3=worsening,4=new).New SLE flare:BILAG 'A' or 'B' event adjudicated to be flare following resolution of entry flare and/or start of prednisone/prednisone-equivalent taper.Inception treatment failure included (entry flare did not subside by Day 57/participant discontinued double-blind period before Day 29).
Time Frame: From start of corticosteroid taper to Day 365
Population: All randomized and treated participants, grouped by the treatment randomized to (ITT).
Measure: Number; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 118 | 57
Participants
  None | 24 | 10
  1 | 47 | 21
  2 | 21 | 10
  >=3 | 17 | 11
  Inception treatment failure | 9 | 5

4. Secondary Outcome: DB; Median Number of Days to the First Occurrence of a New SLE Flare
Description: Elapsed days between start of corticosteroid taper & first day of flare.Scored using BILAG:A:presence of =>1 serious;B:more moderate;C:mild symptomatic;D:prior activity,no current symptoms;E:organ that has never been involved.Calculated based on change during previous 4 weeks (1=improving,2=staying same,3=worsening,4=new).New SLE flare:first BILAG 'A' or 'B' event adjudicated to be flare following resolution of entry flare and/or start of corticosteroid taper.Inception treatment failure included (entry flare did not subside by Day 57/participant discontinued double-blind period before Day 29).
Time Frame: From start of corticosteroid taper to confirmation of disease flare or the end of double-blind period
Population: All randomized and treated participants, grouped by the treatment randomized to (ITT).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 118 | 57
Days | 107.0 [81.0 to 125.0] | 92.0 [58.0 to 150.0]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.7 to 1.5] — Cox proportional-hazards model was used to estimate the hazard ratio of abatacept versus placebo for SLE disease flare. The 95% two-sided confidence interval was provided for the hazard ratio for treatment

5. Secondary Outcome: DB; Number of Participants With a Change in the SLICC/ACR Damage Index at 1 Year Compared to Baseline
Description: SLICC/ACR score or damage index is a measure of cumulative damage due to Systemic Lupus Erythematosus (SLE). Damage is defined as non-reversible change (not related to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months. A score of 0=no damage, early damage is defined as ≥1. The total maximum score is 48, and increasing score indicates increasing disease severity.
Time Frame: From start of study drug treatment to Day 365
Population: All randomized and treated participants who were available for analysis, grouped by the treatment randomized to (ITT).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 107 | 47
participants
  No change | 101 [90.0 to 98.8] | 44 [86.6 to 100.0]
  Increased 1 | 3 [0.6 to 8.0] | 2 [0.5 to 14.5]
  Increased >1 | 3 [0.6 to 8.0] | 1 [0.1 to 11.3]

6. Secondary Outcome: DB; Number of Participants Who Died, Experienced AEs, Other SAEs or Discontinuations Due to AEs, Drug Related AEs
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Drug-related AEs: events with a certain; probable; possible; or missing relationship to the study therapy. Participants who discontinued the study due to an AE were recorded.
Time Frame: Events recorded at each participant encounter, from start of study drug therapy up to Day 337, including up to 56 days after the last dose or up to the first dose of open-label, whichever occurred earlier
Population: All participants given study drug during the double-blind period ("As Treated"). The AEs represented here include SAEs, which are not included in the AE count represented in the AE xml upload section. As such, these numbers may not match.
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 121 | 59
participants
  Deaths | 0 | 0
  AEs | 110 | 54
  SAEs | 24 | 4
  All AEs Leading to Discontinuation | 10 | 3
  Drug related AEs | 59 | 28

7. Secondary Outcome: DB; Number of Participants With Significant AEs of Special Interest
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). For this study, AEs of special interest were associated with the use of immunomodulatory agents. Number of participants with infections, malignant neoplasms, pre-specified autoimmune disorders, acute infusional AEs and peri-infusional AEs were recorded.
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period ("As Treated").Participants grouped for randomized treatments, except where different treatment taken for entire double-blind period (which will instead be presented by first treatment actually received).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 121 | 59
participants
  Infections | 71 | 38
  Malignant neoplasms | 1 | 0
  Pre-specified autoimmune disorders | 4 | 2
  Acute-infusional AEs | 5 | 5
  Peri-infusional AEs | 27 | 13

8. Secondary Outcome: DB; Number of Participants With MAs in Hematology: Hemoglobin, Hematocrit, Erythrocytes and Platelet Count
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Hemoglobin: >3 g/dL decrease from pre-treatment (pre-Rx) value; hematocrit: <0.75* pre-Rx value; erythrocyte count: <0.75* pre-Rx value; platelet count: <0.67* LLN or >1.5* ULN (or, if pre-Rx value <LLN, then <0.5* pre-Rx value or <100000/mm^3).
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period (As Treated) where "not evaluable" was recorded for "high" values (hemoglobin, hematocrit and erythrocytes)has been presented as "0". n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 120 | 58
participants
  Hemoglobin (n = 120, 58) | 1 | 1
  Hematocrit (n=120, 58) | 1 | 1
  Erythrocytes (n=120, 58) | 1 | 1
  Platelet count (n= 118, 58) | 3 | 0

9. Secondary Outcome: DB; Number of Participants With MAs in Hematology: Leukocytes, Neutrophils + Bands (Absolute), Lymphocytes (Absolute), Monocytes (Absolute), Basophils (Absolute) and Eosinophils (Absolute)
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Leukocytes: <0.75* LLN or >1.25* ULN (or, if pre-Rx value <LLN, then <0.8* pre-Rx or >ULN. If pre-Rx value >ULN, then >1.2* pre-Rx or <LLN; Neutrophils+bands (absolute): <1.00* 10^3 cells/microliter (c/uL); Lymphocytes (absolute): <0.75* 10^3 c/uL or >7.50* 10^3 c/uL; Monocytes (absolute): >2000/mm^3; Basophils (absolute): >0.40* 10^3 c/uL; Eosinophils (absolute): >0.75* 10^3 c/uL.
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period ("As Treated") where "not evaluable" was recorded for either "low"(monocytes, basophils and eosinophils) or "high" values(neutrophils)has been presented as "0".n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 120 | 59
participants
  Leukocytes (n = 120, 58) | 26 | 11
  Neutrophils+bands (absolute) (n = 120, 59) | 8 | 2
  Lymphocytes (absolute) (n = 120, 59) | 46 | 30
  Monocytes (absolute) (n = 120, 59) | 1 | 0
  Basophils (absolute) (n = 120, 59) | 0 | 0
  Eosinophils (absolute) (n = 120, 59) | 6 | 2

10. Secondary Outcome: DB: Number of Participants With MAs in Serum Chemistry: ALP, AST, ALT, GGT, Bilirubin (Total), BUN and Creatinine
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria. ALP, GGT: >2* ULN (if pre-Rx >ULN, then >3* pre-Rx); AST, ALT: >3* ULN (if pre-Rx >ULN, then >4* pre-Rx). Bilirubin (total): >2* ULN (if pre-Rx >ULN, then >4* pre-Rx), BUN:>2* pre-Rx; Creatinine:>1.5* pre-Rx.
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period ("As Treated") where "not evaluable" was recorded for "low" values (all parameters) and has been presented as "0". n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 120 | 59
participants
  ALP (n = 120, 59) | 2 | 0
  AST (n = 120, 59) | 3 | 0
  ALT (n = 120, 59) | 2 | 0
  GGT (n = 120, 59) | 3 | 3
  Bilirubin (total) (n = 120, 59) | 0 | 0
  BUN (n = 120, 59) | 4 | 3
  Creatinine (n = 120, 59) | 6 | 4

11. Secondary Outcome: DB; Number of Participants With MAs in Serum Chemistry: Sodium (Serum), Potassium (Serum), Chloride (Serum), Calcium (Total),Protein (Total)
Description: MAs are laboratory measurements marked as abnormal as per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria, Sodium (serum): <0.95* LLN or >1.05* ULN (if pre-Rx <LLN, then <0.95* pre-Rx or >ULN. If pre-Rx >ULN, then >1.05* pre-Rx or <LLN); Potassium (serum), Chloride (serum), protein (total): <0.9* LLN or >1.1* ULN (if pre-Rx <LLN, then <0.9* pre-Rx or >ULN. If pre-Rx >ULN, then >1.1* pre-Rx or <LLN; Calcium (total): <0.8* LLN or >1.2* ULN (if pre-Rx <LLN, then <0.75* pre-Rx or >ULN. If pre-Rx >ULN, then >1.25* pre-Rx or <LLN.
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period ("As Treated").n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 120 | 59
participants
  Sodium (serum) (n = 120, 59) | 1 | 0
  Potassium (serum) (n = 120, 59) | 1 | 1
  Chloride (serum) (n = 120, 59) | 0 | 0
  Calcium (total) (n= 120, 59) | 0 | 0
  Protein (total) (n = 120, 59) | 1 | 0

12. Secondary Outcome: DB; Number of Participants With MAs in Serum Chemistry: Glucose (Serum), Glucose (Fasting Serum), Albumin, Cholesterol (Total), Triglycerides, Fasting Triglycerides
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria, Glucose: <65 mg/dl or >220 mg/dl; Glucose (fasting serum): <0.8* LLN or >1.5 ULN (if pre-Rx <LLN, then <0.8* pre-Rx or >ULN. If pre-Rx >ULN, then >2.0* pre-Rx or <LLN; Albumin: <0.9* LLN (if pre-Rx <LLN, then <0.75 * pre-Rx); cholesterol (total): >2* pre-Rx; triglycerides: >=2.5* ULN, or if pre Rx>ULN then use >2.5* pre Rx; fasting triglycerides: >=2.0* ULN, or if pre Rx>ULN then use >2.0* pre Rx.
Time Frame: as for outcome 6
Population: "All participants given study drug during the double-blind period ("As Treated") where "not evaluable" was recorded for either "low" or "high" values (albumin, cholesterol, triglycerides) has been presented as "0".n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 120 | 59
participants
  Glucose (serum) (n = 120, 59) | 27 | 10
  Glucose, fasting (n = 77, 37) | 5 | 1
  Albumin (n = 120, 59) | 4 | 1
  Cholesterol (total) (n = 118, 58) | 0 | 0
  Triglycerides (n = 75, 36) | 0 | 0
  Triglycerides (fasting) (n = 64, 34) | 0 | 0

13. Secondary Outcome: DB; Number of Participants With MAs in Urinalysis
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following definitions specify the criteria for MAs in urinalysis, Protein, glucose, blood, Leukocyte esterase, RBC, WBC: >=2+ (or, if value >=4, or if pre-Rx value = 0 or 0.5, then >= 2* pre-Rx, or if pre-Rx value =1, then >=3, or if pre-Rx = 2 or 3, then >=4); protein (24 hour urine): >1000 mg/24 hrs and >=2* pre-Rx; GFR: <=60 mL/min/1.73m^2 or > 15% change from baseline; Protein/creatinine ratio: > 100 mg/mmol.
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period ("As Treated") where "not evaluable" was recorded for "low" (protein, glucose, blood, leukocyte esterase, RBC, WBC) or "high" (GFR) values has been presented as "0". n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 120 | 58
participants
  Protein (n = 120, 58) | 15 | 9
  Glucose (n = 120, 58) | 1 | 2
  Blood (n = 120, 58) | 39 | 18
  Leukocyte esterase (n = 107, 51) | 23 | 8
  RBC (n = 107, 55) | 38 | 16
  WBC (n = 115, 54) | 61 | 26
  Protein, 24 hours (n = 89, 40) | 4 | 1
  GFR (n = 120, 59) | 7 | 4
  Protein/creatinine ratio (n = 119, 58) | 11 | 4

14. Secondary Outcome: DB; Number of Participants With Clinically Significant Abnormal Vital Signs and/or Physical Examination Findings
Description: Vital signs assessments and physical examination were conducted throughout the study. Vital signs assessments included body temperature, respiratory rate, blood pressure (systolic and diastolic) and heart rate. The investigator used his/her clinical judgment to decide whether or not abnormalities in vital signs or physical examination were clinically meaningful.
Time Frame: as for outcome 6
Population: All participants given study drug during the double-blind period ("As Treated"). Significant vital signs and physical examination findings are reported in the AE tables. Symptoms related to lupus were collected in British Isles Lupus Assessment Group (BILAG) assessments.
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Open Label Period (OL); Number of Participants Who Died, Experienced Adverse Events (AEs), Serious AEs, Drug Related AEs or SAEs and Discontinued Due to AEs
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to an AE were recorded. Drug-related AEs or SAEs: events with a relationship to the study therapy of certain; probable; possible; or missing.
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: As treated analysis population: All treated participants who entered the open-label period and received at least one dose of study medication during open-label period.
Measure: Number; unit: participants
Groups:
- Abatacept: Participants were administered with abatacept (10mg/kg) iv infusion over approximately 30 minutes on Days 365, 393, 421 and every 28 days thereafter up to and including Day 729. All participants received a dose based on their screening visit weight (participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg and participants weighing > 100 kg received 1000mg).
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Deaths | 1
  AEs | 97
  SAEs | 21
  All AEs Leading to Discontinuation | 3
  Drug related AEs | 49
  Drug related SAEs | 11

16. Primary Outcome: OL; Number of Participants With Significant AEs of Special Interest
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). For this study, it was decided that AEs of particular importance were associated with the use of immunomodulatory agents. Number of participants with infections, malignant Neoplasms, pre-specified autoimmune disorders, acute-infusional AEs and peri-infusional AEs were recorded.
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Infections | 82
  Malignant neoplasms | 1
  Pre-specified autoimmune disorders | 4
  Acute-infusional AEs | 3
  Peri-infusional AEs | 15

17. Primary Outcome: OL; Number of Participants With Marked Abnormalities (MAs) in Hematology: Hemoglobin, Hematocrit, Erythrocytes and Platelet Count
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Hemoglobin: >3 g/dL decrease from pre-treatment (pre-Rx) value; hematocrit: <0.75* pre-Rx value; erythrocyte count: <0.75* pre-Rx value; platelet count: <0.67* lower limit of normal (LLN) or >1.5* upper limit of normal (ULN) (or, if pre-Rx value <LLN, then <0.5* pre-Rx value or <100000/mm^3).
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: As treated analysis population: All treated participants who entered the open-label period and received at least one dose of study medication. Where "not evaluable" was recorded for "high" values (hemoglobin, hematocrit, erythrocytes) and has been presented as "0". n = number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Hemoglobin (n = 110) | 2
  Hematocrit (n = 110) | 3
  Erythrocytes (n = 110) | 2
  Platelet count (n = 108) | 3

18. Primary Outcome: OL; Number of Participants With MAs in Hematology: Leukocytes, Neutrophils + Bands (Absolute), Lymphocytes (Absolute), Monocytes (Absolute), Basophils (Absolute) and Eosinophils (Absolute)
Description: MMAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Leukocytes: <0.75* LLN or >1.25* ULN (or, if pre-Rx value <LLN, then <0.8* pre-Rx or >ULN. If pre-Rx value >ULN, then >1.2* pre-Rx or <LLN; Neutrophils+bands (absolute): <1.00* 10^3 cells/microliter (c/uL); Lymphocytes (absolute): <0.75* 10^3 c/uL or >7.50* 10^3 c/uL; Monocytes (absolute): >2000/mm^3; Basophils (absolute): >0.40* 10^3 c/uL; Eosinophils (absolute): >0.75* 10^3 c/uL.
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: As treated analysis population: All treated participants who entered the open-label period and received at least one dose of study medication during open-label period. Where "not evaluable" was recorded for either "low"(monocytes, basophils, eosinophils) or "high"(neutrophils) has been presented as "0".
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Leukocytes | 18
  Neutrophils+bands (absolute) | 6
  Lymphocytes (absolute) | 32
  Monocytes (absolute) | 0
  Basophils (absolute) | 0
  Eosinophils (absolute) | 3

19. Primary Outcome: OL; Number of Participants With MAs in Serum Chemistry: Alkaline Phosphatase (ALP), Aspartate-aminotransferase (AST), Alanine-aminotransferase (ALT), Gamma-glutamyl Transferase (GGT), Bilirubin(Total), Blood Urea Nitrogen (BUN), Creatinine
Description: as for outcome 10
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: As treated analysis population: All treated participants who entered the open-label period and received at least one dose of study medication during open-label period. Where "not evaluable" was recorded for "low" values (ALP, AST, ALT, GGT, bilirubin, BUN, creatinine) and has been presented as "0".
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  ALP | 0
  AST | 3
  ALT | 4
  GGT | 6
  Bilirubin (total) | 0
  BUN | 3
  Creatinine | 7

20. Primary Outcome: OL; Number of Participants With MAs in Serum Chemistry: Sodium (Serum), Potassium (Serum), Chloride (Serum), Calcium (Total), Protein (Total)
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria, Sodium (serum): <0.95x LLN or >1.05x ULN (if pre-Rx<LLN, then <0.95x pre-Rx or >ULN. If pre-Rx >ULN, then >1.05x pre-Rx or <LLN); Potassium (serum), Chloride (serum), protein (total): <0.9x LLN or >1.1xULN (if pre-Rx <LLN, then <0.9xpre-Rx or >ULN. If pre-Rx >ULN, then >1.1xpre-Rx or <LLN; Calcium (total): <0.8xLLN or >1.2xULN (if pre-Rx <LLN, then <0.75x pre-Rx or >ULN. If pre-Rx >ULN, then >1.25x pre-Rx or <LLN.
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Sodium (serum) | 0
  Potassium (serum) | 7
  Chloride (serum) | 0
  Calcium (total) | 1
  Protein (total) | 4

21. Primary Outcome: OL; Number of Participants With MAs in Serum Chemistry: Glucose (Serum), Glucose (Fasting Serum), Albumin, Cholesterol (Total), Triglycerides, Fasting Triglycerides
Description: MAs are laboratory measurements marked as abnormal, as per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria, Glucose: <65 mg/dL or >220 mg/dL; Glucose (fasting serum): <0.8* LLN or >1.5 ULN (if pre-Rx <LLN, then <0.8* pre-Rx or >ULN. If pre-Rx >ULN, then >2.0* pre-Rx or <LLN; Albumin: <0.9* LLN (if pre-Rx <LLN, then <0.75 * pre-Rx); cholesterol (total): >2* pre-Rx; triglycerides: >=2.5* ULN, or if pre Rx>ULN then use >2.5* pre Rx; fasting triglycerides: >=2.0* ULN, or if pre Rx>ULN then use >2.0* pre Rx.
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: As treated analysis population: All treated participants who entered the open-label period and received at least one dose of study medication. Where "not evaluable" was recorded for either "low" (cholesterol, triglycerides) or "high" (albumin) has been presented as "0". n = number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Glucose (serum) (n = 110) | 21
  Glucose (fasting serum) (n = 55) | 6
  Albumin (n = 110) | 6
  Cholesterol (total) (n = 15) | 0
  Triglycerides (n = 10) | 0
  Triglycerides (fasting) (n = 9) | 0

22. Primary Outcome: OL; Number of Participants With MAs in Urinalysis
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following definitions specify the criteria for MAs in urinalysis, Protein, glucose, blood, Leukocyte esterase, red blood cells (RBC), white blood cells (WBC): >=2+ (or, if value >=4, or if pre-Rx value = 0 or 0.5, then >= 2* or if pre-Rx value =1, then >=3, or if pre-Rx = 2 or 3, then >=4); protein (24 hour urine): >1000 mg/24 hrs and >=2* pre-Rx; Glomerular filtration rate (GFR): <=60 mL/min/1.73m^2 or > 15% change from baseline; Protein/creatinine ratio: > 100 mg/mmol.
Time Frame: From start of study drug therapy in open-label period (Day 365) up to 56 days after the last dose of open-label period
Population: As treated analysis population: all treated participants who entered the OL period and received at least 1 dose of study medication. Where "not evaluable" was recorded for "low" (protein, glucose, blood, leukocyte esterase, RBC, WBC) or "high"(GFR) values and presented as "0". n=number of participants with evaluable results (each arm respectively).
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 110
participants
  Protein (n = 110) | 12
  Glucose (n= 110) | 0
  Blood (n = 110) | 41
  Leukocyte esterase (n = 104) | 28
  WBC (n = 105) | 57
  RBC (n = 101) | 35
  GFR (n = 110) | 9
  Protein/creatinine ratio (n = 109) | 10

23. Secondary Outcome: DB; Number of Participants With Antibodies Specific for CTLA4-T and Abatacept, Following Abatacept Treatment
Description: Electrochemiluminescence (ECL) immunoassay based on Meso Scale Discovery (MSD) technology was used to detect antibodies specific for CTLA4-T and for abatacept.
Time Frame: From Day 1 to Day 365
Population: Participants who received abatacept and for whom baseline and at least one additional measurement during double-blind period were available.
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 121
participants | 2

24. Secondary Outcome: OL; Number of Participants With a New SLE Flare
Description: SLE flares scored using BILAG:A:presence of =>1 serious lupus features;B:more moderate features;C:mild symptomatic features;D:prior activity with no current symptoms due to active lupus;E:an organ that has never been involved.BILAG scores based on degrees of change in clinical features (1=improving,2=staying the same,3=worsening,4=new).New SLE flare means new BILAG A/B features in any organ system.Based on the recommendation of the Data Monitoring Committee, open-label period terminated, as failed to meet primary outcome measure for double-blind period/increase in SAEs in abatacept group.
Time Frame: From start of study drug therapy in open-label period (Day 365), Day 393, 421, 449 and every 28 days thereafter till Day 729.
Population: as for outcome 15
Arm/Group | Abatacept
Number analyzed (Participants) | 0

25. Secondary Outcome: OL; Number of Participants With a Change in the SLICC/ACR Damage Index at Year 2 Compared to Baseline
Description: SLICC/ACR damage index:measure of cumulative damage due to SLE.Damage=non-reversible change occurring since onset of lupus,ascertained by clinical assessment & present for =>6 months.Scores of SLICC/ACR index:1:single episode;2:repeated episodes at least 6 months apart.Change in score from baseline to 1 year presented as:no change,increase 1 (an increase in score of 1),increase >1 (an increase in score of >1).Based on recommendation of Data Monitoring Committee, open-label period terminated, as failed to meet primary outcome measure for double-blind period/increase in SAEs in abatacept group.
Time Frame: From start of study drug therapy in open-label period (Day 365) and on Day 729.
Population: as for outcome 15
Arm/Group | Abatacept
Number analyzed (Participants) | 0

26. Secondary Outcome: OL; Total Number of BILAG A Flares Each Participant Experienced
Description: Total number of BILAG A flares in any organ system after steroid tapering = new BILAG A features in any organ system. Scores defined as follows: None: participants with no BILAG A flare; 1: participants with 1 BILAG A flare or participants who discontinued without a new BILAG A flare were imputed as having one event. 2: participants with 2 BILAG A flares; 3 or >3: participants with 3 or more BILAG A flares.Based on recommendation of Data Monitoring Committee, open-label period terminated, as failed to meet primary outcome measure for double-blind period/increase in SAEs in abatacept group.
Time Frame: as for outcome 24
Population: as for outcome 15
Groups:
- Abatacept: Participants were administered intravenous (iv) infusions of abatacept (10 mg/kg) over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 337. All participants received a dose based on their screening visit weight (participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg and participants weighing > 100 kg received 1000mg). Prednisone or prednisone equivalent was administered at an initial oral dose of 30 mg once daily (OD). A standardized prednisone or prednisone equivalent taper procedure was followed whenever the participant's clinical features qualified for British Isles Lupus Assessment Group (BILAG) "C" or "D" status after Day 29. BILAG A: presence of one or more serious features of lupus; BILAG B: more moderate features of the disease; BILAG C: mild symptomatic features; BILAG D: prior activity with no current symptoms due to active lupus; BILAG E: an organ that has never been involved.
Arm/Group | Abatacept
Number analyzed (Participants) | 0

27. Secondary Outcome: OL; Area Under the Curve (AUC) for Prednisone or Prednisone Equivalent
Description: Total exposure to glucocorticosteroid was measured by the total prednisone or prednisone equivalent AUC. Based on the recommendation of the Data Monitoring Committee, the open-label, long-term extension period was terminated by the sponsor, for failure to meet the primary outcome measure for the double-blind period and because of an increase in SAEs in the abatacept treatment group. As such, these data were not analyzed.
Time Frame: as for outcome 24
Population: as for outcome 15
Arm/Group | Abatacept
Number analyzed (Participants) | 0

28. Secondary Outcome: OL; Number of Participants With Antibodies Specific for CTLA4-T and Abatacept, Following Abatacept Treatment
Description: MSD technology was used to detect antibodies specific for CTLA4-T and for abatacept.
Time Frame: After the first dose of open-label period
Population: Immunogenicity analysis population: participants who received abatacept and for whom baseline and at least one additional measurement during the open-label period were available.
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 108
participants | 30

ADVERSE EVENTS:
Time Frame: Events recorded at each participant encounter, from start of study drug therapy up to Day 337, including up to 56 days after the last dose or up to the first dose of open-label, whichever occurred earlier.
Groups:
- Abatacept: Participants were administered abatacept (10 mg/kg) IV over approximately 30 minutes on Days 1, 15, 29 and every 28 days thereafter up to and including Day 337. All participants received a dose based on screening visit weight. Prednisone or prednisone equivalent was administered at an initial oral dose of 30 mg once daily (OD). A standardized prednisone or prednisone equivalent taper procedure was followed whenever the participant's clinical features qualified for British Isles Lupus Assessment Group (BILAG) "C" or "D" status after Day 29. Participants who completed the double-blind period were eligible for the open-label long-term extension period, where all participants were reallocated to abatacept (regardless of randomized treatment in the double-blind period) according to body weight at study entry. Infusions continued every 28 days until abatacept was marketed for SLE or the drug development program discontinued.
Arm/Group | Abatacept | Placebo
Serious Adverse Events (participants affected / at risk) | 24/121 | 4/59
Other Adverse Events (participants affected / at risk) | 90/121 | 41/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=121) | Placebo (N=59)
PERICARDITIS (Cardiac disorders) | 2 | 0
LUPUS VASCULITIS (Vascular disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 1 | 0
ACUTE POLYNEUROPATHY (Nervous system disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
PERITONITIS LUPUS (Gastrointestinal disorders) | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1
LUPUS NEPHRITIS (Renal and urinary disorders) | 1 | 0
GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0
MESANGIOPROLIFERATIVE GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 3 | 1
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PYREXIA (General disorders) | 3 | 0
CHEST PAIN (General disorders) | 1 | 0
FACE OEDEMA (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=121) | Placebo (N=59)
PALPITATIONS (Cardiac disorders) | 2 | 4
HYPERTENSION (Vascular disorders) | 4 | 3
INSOMNIA (Psychiatric disorders) | 10 | 5
DEPRESSION (Psychiatric disorders) | 7 | 3
HEADACHE (Nervous system disorders) | 25 | 10
DIZZINESS (Nervous system disorders) | 6 | 5
NAUSEA (Gastrointestinal disorders) | 12 | 4
DIARRHOEA (Gastrointestinal disorders) | 14 | 4
CONSTIPATION (Gastrointestinal disorders) | 2 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 5
INFLUENZA (Infections and infestations) | 7 | 3
SINUSITIS (Infections and infestations) | 8 | 4
BRONCHITIS (Infections and infestations) | 7 | 4
PHARYNGITIS (Infections and infestations) | 3 | 4
GASTROENTERITIS (Infections and infestations) | 7 | 2
NASOPHARYNGITIS (Infections and infestations) | 3 | 7
URINARY TRACT INFECTION (Infections and infestations) | 13 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 25 | 9
ACNE (Skin and subcutaneous tissue disorders) | 7 | 0
RASH (Skin and subcutaneous tissue disorders) | 4 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 5
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 3
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 | 2
CHEST PAIN (General disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.